## Tailoring Surgical Management of Multifocal Breast Cancer:is There a Possibility

## NCT03900299

**Document Date: December 2, 2019** 

## **Data Management and Analysis:**

The collected data was revised, coded, tabulated and introduced to a PC using Statistical package for Social Science ((IBM Corp. Released 2011. IBM SPSS Statistics for Windows, Version 20.0. Armonk, NY: IBM Corp). Data was presented and suitable analysis was done according to the type of data obtained for each parameter as follow:

I-Descriptive statistics:-Frequency and percentage of qualitative variables.

## **II-Analytical statistics:**

- 1. Chi-Square test was used to examine the relationship between two qualitative variables
- **2. Fisher's exact test:** was used to examine the relationship between two qualitative variables for 2x2 tables (tables with 4 cells), when the expected count is less than 5 in more than 20% of cells
- 3-Monte Carlo-test was used to examine the relationship between two qualitative variables for larger than 2x2 tables (tables with more than 4 cells) when the expected count is less than 5 in more than 20% of cells
  - P- value: level of significance

-P>0.05: Non significant (NS).

-P< 0.05: Significant (S).

-P<0.01: Highly significant (HS).